CLINICAL TRIAL: NCT01353846
Title: Comparison Between Natural and Artificial Cycle in Recipient Oocyte Patients
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Instituto Valenciano de Infertilidad, IVI VALENCIA (Other)
Responsible Party: Dra. Pilar Alamá, IVI Valencia
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 0901-C-055-MF
Record Dates: First submitted 2011-05-10; First posted 2011-05-16 (Estimated); Last update posted 2012-04-02 (Estimated); Status verified 2012-03

CONDITIONS: Infertility
Keywords: oocyte donation program; natural cycle; hormone replacement therapy
MeSH Terms: conditions — Infertility | interventions — Control Groups; Estradiol; Progesterone; Triptorelin Pamoate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Natural cycle (Active Comparator)
  Interventions: Other: observation natural cycle
- Artificial cycle (Active Comparator): Drugs: Agonist GnRH Acetate Triptoreline Acetate Triptorelina (Agonist GnRH), 3.75 mg. single dose. Estradiol Valerate, orally Initially 4 pills daily during 4 days, and after increase the dose to 6 mg orally daily.
  Natural micronized progesterone, 400 mg/12 hours vaginal administration
  Interventions: Drug: Agonist GnRH; estradiol Valerate; progesterone

INTERVENTIONS:
Other: observation natural cycle — The patients natural reproductive cycle will be observed and compared to the second arm.
  Other Names: Control group with natural menstration cycle.
  Arms: Natural cycle
Drug: Agonist GnRH; estradiol Valerate; progesterone — Medications: Agonist GnRH Acetate Triptoreline and Acetate Triptorelina and Estradiol Valerate and Natural micronized progesterone, 400 mg/12 hours vaginal administration
  Other Names: Decapeptyl (IPSEN)3.75 mg.; Progynova 1 mg (Bayer Schering Farma); Natural micronized progesterone 400 mg/12 hours
  Arms: Artificial cycle

SUMMARY:
The purpose of this study is to compare the natural cycle (without any medication) with the well-established artificial cycle in an egg donation program.

DETAILED DESCRIPTION:
Oocyte donation is an assisted reproduction technique well established. In patients with ovarian function, it is necessary to synchronize the cycle of the egg donor with the recipient, usually through endometrial preparation of the recipient by artificial cycle, by administering a GnRH agonist on day 21 of cycle and then administered increasing doses of estrogen therapy to achieve adequate endometrial thickness.

The necessity of synchronization between donors and recipient, has made possible not routinely the natural cycle for oocyte donation.

The investigators have recently introduced oocyte vitrification and it allows us to plan the egg donation in a different way. Now the investigators can previously cryopreserved donor oocytes and at the time that the investigators have a compatible receiver, then, plan the donation In this study it will be possible compare the results of oocyte donation cycles in terms of pregnancy rate, implantation and liveborn, depending on whether the recipient has made an artificial cycle of preparation endometrial or a natural cycle.

ELIGIBILITY:
Inclusion Criteria:

* infertile females with preserved gonadal function
* ages 18 - 44 years old included
* first oocyte donation cycle

Exclusion Criteria:

* BMI: > 28
* recurrent miscarriages (3 or more)
* recurrent of implantation failure
* severe male factor
* important miomas
* > 44 years old
* Problems with the drugs used in the study

Ages: 18 Years to 44 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 70 (Estimated)
Dates: Start 2011-05; Primary Completion 2012-11 (Estimated); Study Completion 2012-11 (Estimated)

PRIMARY OUTCOMES:
Preparation and treatment for Assisted Human Reproduction procedures and in the case opf pregnancy, follow up. | 12 months
  Outcome of the study is measured by the pregnancy rates after IVF treatments of both arms.

CONTACTS AND LOCATIONS:
Overall Officials: Dra. Pilar Alamá, MDPhD, Study Director — IVI Valencia
Locations (1):
- IVI Valencia, Valencia, Valencia, Spain